CLINICAL TRIAL: NCT04027686
Title: Clinical Evaluation of WaterLase (iPlus) Laser Therapy Used as an Adjunct to Non-Surgical Treatment of Chronic Periodontitis: A Randomized, Controlled, Split-Mouth Clinical Study
Brief Title: Clinical Evaluation of Laser Therapy Used as an Adjunct to Non-Surgical Treatment of Gum Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Biolase Inc (Industry)
Responsible Party: Principal Investigator, Perry R Klokkevold, DDS, MS, Professor of Clinical Dentistry, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB#15-000519
Record Dates: First submitted 2019-07-18; First posted 2019-07-22 (Actual); Results first posted 2021-03-05 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-02

CONDITIONS: Periodontitis Chronic Generalized Moderate; Periodontitis Chronic Generalized Severe
Keywords: Laser Therapy; Non-surgical periodontal therapy; Scaling and root planing
MeSH Terms: interventions — Laser Therapy; Root Planing

STUDY DESIGN:
Intervention Model Description: Randomized, Controlled, Split-mouth
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- SRP + Adjunctive Laser Therapy (Experimental): Laser therapy used as an adjunct to scaling and root planing
  Interventions: Device: Laser Therapy; Procedure: Non-surgical Scaling and Root Planing
- SRP alone (Active Comparator): Scaling and root planing used as conventional non-surgical periodontal therapy
  Interventions: Procedure: Non-surgical Scaling and Root Planing

INTERVENTIONS:
Device: Laser Therapy — Adjunctive application of laser therapy in the periodontal pocket
  Arms: SRP + Adjunctive Laser Therapy
Procedure: Non-surgical Scaling and Root Planing — Scaling to remove calculus deposits and root planing to smooth root surfaces

SUMMARY:
The use of lasers to treat various problems in dentistry is growing as it has in medicine. One application is the use of lasers to treat periodontal disease. It has been suggested that the laser may reduce the need for surgical treatment by reducing pockets. The goal of this study is to evaluate the effectiveness of laser treatment for periodontal disease. Laser therapy will be used in addition to traditional non-surgical scaling and root planing (deep cleaning). The information obtained from this study will provide an objective assessment of adjunctive laser therapy compared to conventional periodontal therapy and will attempt to show the benefits, if any, lasers can provide in the treatment of chronic periodontal disease.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years old or older (male or female)
* Healthy without systemic diseases that may adversely effect healing
* Not pregnant and no current plans to become pregnant
* No periodontal treatment in the previous 12 months
* No systemic antibiotic therapy in the previous 6 months
* At least two quadrants with periodontitis (ideally opposite side same jaw)
* Each quadrant must have two or more sites with probing pocket depths ≥ 5mm
* Each quadrant should include interproximal intrabony defect(s)

Exclusion criteria:

* Any systemic disease, medication, or habit known to adversely influence bone metabolism and/or wound healing:
* Poorly controlled diabetes (HbA1c > 7%)
* History of bisphosphonate medications
* History of radiation therapy affecting the proposed treatment site(s)
* History of immunosuppressive medications (e.g. corticosteroids)
* History of tobacco use (current or past tobacco use within the past 1 year)
* Immune compromise caused by disease, treatment or other condition
* Recent history of periodontal surgery (within the previous 2 years)
* Recent history of scaling and root planing (within the previous 12 months)
* Any condition that contraindicates periodontal therapy including surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Perry R Klokkevold, DDS, MS, Principal Investigator — UCLA School of Dentistry, Section of Periodontics

RESULTS

PARTICIPANT FLOW:
Groups:
- Periodontal Sites Assigned to SRP or SRP + Adjunctive Laser Therapy: Each participant had one or more periodontal sites randomly assigned to scaling and root planing only (Standard of Care) or to Laser therapy in addition to scaling and root planing
- Pilot Procedure Arm: Preliminary enrollment of individuals to pilot-test the protocol
Period: Overall Study
Arm/Group | Periodontal Sites Assigned to SRP or SRP + Adjunctive Laser Therapy | Pilot Procedure Arm
Started | 17 | 6
Completed | 15 | 5
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 2 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: 17 participants were enrolled in the main study, with a total of 49 Test and 49 Control sites (periodontal pockets)
Groups:
- Periodontal Sites Assigned to SRP + Adjunctive Laser Therapy or SRP Alone: Enrolled participants each had multiple periodontal sites randomly assigned to receive scaling and root planing as conventional non-surgical periodontal therapy, or Laser therapy as an adjunct to scaling and root planing.
- Total: Total of all reporting groups
Arm/Group | Periodontal Sites Assigned to SRP + Adjunctive Laser Therapy or SRP Alone | Pilot Procedure Arm | Total
Number analyzed (Participants) | 17 | 6 | 23
Age, Categorical [Count of Participants; unit: Participants] — Population: Each participant was treated with both SRP + Adjunctive Laser Therapy (test) and SRP alone (control) in separate quadrants. Thus, the total number of participants is the same number observed in each group. Subjects served as their own control.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 16 | 6 | 22
    >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 2 | 14
  Male | 5 | 4 | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 17 | 6 | 17

OUTCOME MEASURES:

1. Primary Outcome: Probing Pocket Depth
Description: This is a measure from base of pocket to gingival margin.
Time Frame: 12 months
Population: 15 participants had a total of 90 periodontal pockets, randomized 45 to Test and 45 to Control interventions. Each site had one buccal and one lingual measurement, with measures < 4mm excluded from analyses. The preliminary pilot participants were not assessed for outcome measures.
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Periodontal pockets
Arm/Group | SRP + Adjunctive Laser Therapy | SRP Alone | Pilot Procedure Arm
Number analyzed (Participants) | 15 | 15 | 0
Number analyzed (Periodontal pockets) | 78 | 77 | 0
mm | 4.167 (0.986) | 4.273 (1.232) |

2. Primary Outcome: Sites That Bleed on Probing
Description: Percentage of sites that bleed in response to probing. Bleeding observed within 30 seconds from pocket/sulcus following periodontal probe measurement.
Time Frame: 12 months
Population: 15 participants had a total of 90 periodontal pockets, randomized 45 to Test and 45 to Control interventions. Each site had one buccal and one lingual measurement, with measures <4mm excluded from analyses. Pilot enrollees were not assessed for outcome measures.
Measure: Number; unit: percentage of sites with bleeding
Units Other Than Participants: Periodontal pockets
Arm/Group | SRP + Adjunctive Laser Therapy | SRP Alone | Pilot Procedure Arm
Number analyzed (Participants) | 15 | 15 | 0
Number analyzed (Periodontal pockets) | 78 | 77 | 0
percentage of sites with bleeding | 55.1 | 63.6 |

3. Primary Outcome: Gingival Recession
Description: Measure of gingival recession following treatment. This is a measure of the gingival margin from the cement-enamel junction.
Time Frame: 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Periodontal pockets
Arm/Group | SRP + Adjunctive Laser Therapy | SRP Alone | Pilot Procedure Arm
Number analyzed (Participants) | 15 | 15 | 0
Number analyzed (Periodontal pockets) | 78 | 77 | 0
mm | 1.167 (1.263) | 1.182 (1.305) |

4. Primary Outcome: Clinical Attachment Level
Description: Periodontal clinical attachment level following treatment. This is a calculation (clinical attachment level = probing pocket depth + gingival recession).
Time Frame: 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Periodontal pockets
Arm/Group | SRP + Adjunctive Laser Therapy | SRP Alone | Pilot Procedure Arm
Number analyzed (Participants) | 15 | 15 | 0
Number analyzed (Periodontal pockets) | 78 | 77 | 0
mm | 5.346 (1.578) | 5.455 (1.766) |

5. Secondary Outcome: Periodontal Microbiome
Description: Assess changes in periodontal microbiome using DNA sequencing
Time Frame: 12 months
Population: Microbiome results will not be available for analysis until April 2021
Arm/Group | SRP + Adjunctive Laser Therapy | SRP Alone
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Patient Reported Outcomes: VAS Questionnaire
Description: Measure patient reported pain (0-100), comfort (0-100), sensitivity (0-100) and satisfaction (0-100) using VAS questionnaire, with lower values indicating better outcome for pain and sensitivity and higher values indicating better outcome for comfort and satisfaction.
Time Frame: 12 months
Population: 15 participants had a total of 90 sites (periodontal pockets), randomized 45 to Test and 45 to Control interventions. Pilot enrollees were not assessed for outcome measures.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Periodontal pocket sites
Arm/Group | SRP + Adjunctive Laser Therapy | SRP Alone | Pilot Procedure Arm
Number analyzed (Participants) | 15 | 15 | 0
Number analyzed (Periodontal pocket sites) | 45 | 45 | 0
units on a scale
  Pain | 2.316 (6.634) | 1.056 (3.334) |
  Comfort | 100 (0) | 100 (0) |
  Sensitivity | 16.158 (30.848) | 20.833 (32.787) |
  Satisfaction | 99.579 (1.853) | 99.611 (1.65) |

ADVERSE EVENTS:
Time Frame: 12 months
Groups:
- SRP + Adjunctive Laser Therapy: Laser therapy used as an adjunct to scaling and root planing
  Following patient identification, review of health history and checking vital signs, local anesthesia is applied to the area.
  Laser Therapy: Adjunctive application of laser therapy to de-epithelialize the outer surface of gingival margin and within the periodontal pocket. The inner pocket epithelium is removed from the free gingival margin to the level equal with the pocket depth.
  Non-surgical Scaling and Root Planing: Scaling with ultrasonic scaler and hand instruments to remove calculus deposits and root planing to smooth root surfaces.
  Laser Therapy: Following non-surgical scaling and root planing, laser is used to remove smear layer from root surface, to completely remove pocket lining and to degranulate the pocket. Laser is used to decorticate and stimulate the bone at the base of defect. Finally, the laser is used to remove the residual debris while inducing blood coagulation.
  The surgical site is compressed with moistened 2 x 2 gauze using finger pressure for several minutes to achieve hemostasis.
- SRP Alone: Scaling and root planing used as conventional non-surgical periodontal therapy
  Following patient identification, review of health history and checking vital signs, local anesthesia is applied to the area.
  Non-surgical Scaling and Root Planing: Scaling with ultrasonic scaler and hand instruments to remove calculus deposits and root planing to smooth root surfaces. Pockets were flushed with ultrasonic scaler.
Arm/Group | SRP + Adjunctive Laser Therapy | SRP Alone | Pilot Procedure Arm
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/17 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17 | 0/5
Other Adverse Events (participants affected / at risk) | 0/17 | 0/17 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-30): https://cdn.clinicaltrials.gov/large-docs/86/NCT04027686/Prot_SAP_000.pdf